CLINICAL TRIAL: NCT06429215
Title: Preventing Cognitive Decline and Dementia Through an Innovative Immersive Virtual Reality and Telemedicine-based Multi-component Intervention: a Randomized Controlled Trial
Brief Title: REducing the Risk of COgnitive DEcline ad Dementia in Patients With Subjective Cognitive Decline Through an Immersive Virtual Reality and Telemedicine-based Multi-component Intervention: the SCD-ReCODED Study
Acronym: SCD-ReCODED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Maria Stefania De Simone, Principal investigator, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRIN 2022 PNRR P2022E3CZY
Record Dates: First submitted 2024-05-10; First posted 2024-05-24 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Subjective Cognitive Decline
Keywords: Subjective cognitive decline; Multi-component training; Non-pharmacological intervention; Virtual reality; Telemedicine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multi-component Intervention (MC-I) (Experimental): VR cognitive training + Psychoeducation program
  Interventions: Device: Multi-component Intervention (MC-I): VR Cognitive training and Psychoeducation on health and lifestyle
- Cognitive-only intervention (CO-I) (Active Comparator): VR Cognitive training + Psychoeducation active control
  Interventions: Device: Cognitive-only intervention (CO-I): VR Cognitive training (+ Psychoeducation active control)
- Active control intervention (AC-I) (Active Comparator): VR Cognitive active control + Psychoeducation active control
  Interventions: Device: Active control intervention (AC-I): VR Cognitive active control + Psychoeducation active control

INTERVENTIONS:
Device: Multi-component Intervention (MC-I): VR Cognitive training and Psychoeducation on health and lifestyle — In a period of 5 consecutive weeks, participants will receive:
  * an interactive immersive virtual reality cognitive training for 30 minutes, 3 days per week. It consists in different tasks implemented in virtual real-like scenarios of daily living situations that target the following cognitive processes: long-term associative memory, relational binding, spatial pattern separation and pattern completion;
  * an interactive immersive virtual reality health and lifestyle education program for 30 minutes, 1 day per week. It consists in 360° videos aimed at advancing awareness and knowledge of the various health conditions associated with an increased risk of cognitive decline and dementia and helping participants to develop a healthier lifestyle.
  Arms: Multi-component Intervention (MC-I)
Device: Cognitive-only intervention (CO-I): VR Cognitive training (+ Psychoeducation active control) — In a period of 5 consecutive weeks, participants will receive:
  * the interactive immersive virtual reality cognitive training as described in the MC-I condition, for about 30 minutes, 3 days per week;
  * an active control of the immersive virtual reality psychoeducation program for 30 minutes, 1 day per week.
  Arms: Cognitive-only intervention (CO-I)
Device: Active control intervention (AC-I): VR Cognitive active control + Psychoeducation active control — In a period of 5 consecutive weeks, participants will receive:
  * an active control of the immersive virtual reality cognitive training (participants will be requested to virtually carry out daily actions, in the same setting as those performed in cognitive immersive VR training, but they will follow prearranged instructions requiring very low cognitive demands) for about 30 minutes, 3 days per week;
  * an active control of the immersive virtual reality psychoeducation program for about 30 minutes, 1 day per week.
  Arms: Active control intervention (AC-I)

SUMMARY:
Older adults with subjective cognitive decline (SCD) are at high risk of developing dementia and frequently experience subclinical symptoms (e.g., anxiety, depression) which are themselves associated with dementia and cognitive decline risk. To date, the lack of effective disease-modifying treatments, along with the reliable identification of modifiable lifestyle risk factors (e.g., cognitive activity, dietary habits, physical exercise), have led to growing interest to invest in non-pharmacological interventions that may reduce the prevalence and incidence of dementia and cognitive decline in older adults. In this framework, the aim of this project is to evaluate the efficacy of an Immersive Virtual Reality (IVR) and telemedicine-based multi-component intervention, combining cognitive training and a health and lifestyle education program, for preventing cognitive decline and dementia in at-risk individuals (i.e., SCD). For this purpose, a randomized, double-blinded controlled trial (RCT) will be conducted on seventy-five eligible individuals with SCD, who will be randomly assigned to one of three conditions: (a) multi-component intervention (MC-I), including SCD-tailored cognitive IVR training plus a health and lifestyle education program, (b) cognitive-only intervention (CO-I), including the SCD-tailored cognitive IVR training plus an active control for the education program, and (c) active control intervention (AC-I) for both cognitive training and education program. Intervention will be provided in 20 at-home sessions (4 sessions/week, each lasting about 30 minutes) over a period of 5 weeks. Outcome measures include clinical, neuropsychological, behavioural and neuroimaging data that will be collected before and immediately after intervention in order to detect potentially intervention-induced changes in objective cognitive functioning (primary outcome), subjective cognitive functioning, mood, quality of life and brain connectivity (secondary outcome). Users' compliance with IVR and telemedicine approach will be also evaluated, as well as individuals' factors affecting training efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Self-perceived decline in cognition compared to five years ago
* Lack of objective cognitive impairment.

Exclusion Criteria:

* Clinically significant depression and anxiety;
* Psychiatric disorders;
* Unstable medical conditions.
* Severe visual, auditory, verbal or physical impairments interfere with communication, command compliance, and strategy execution
* Dizziness or epilepsy history;

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive functioning (1): change scores on the Face-Name Associative Memory Exam | Baseline, post-intervention (around 6 weeks after baseline)
  The Face-Name Associative Memory Exam (short form - FNAME12) is an associative long-term memory task that requires the participant to learn and retrieve 12 novel face-name and face-occupation pairs. It consists of two learning phases, followed by an immediate cued recall and a 30-min delayed recall and recognition trial. For each trial, scores range from 0 to 12, where higher scores indicate better memory performance.
Cognitive functioning (2): change scores on the Visual Short-Term Memory Binding Test | Baseline, post-intervention (around 6 weeks after baseline)
  The Visual Short-Term Memory Binding Test is a recognition task based on a change detection paradigm for arrays of stimuli presented on a computer screen. Two conditions are investigated, that is, a shape-only condition as the first and a shape-color condition as the second. In both conditions, participants are asked to remember visual arrays of two or three black polygons (in the shape-only condition) or colored polygons (in the shape-color condition) presented for 2 s (study phase). For each condition, scores range from 0 to 32, where higher scores indicate better memory performance.
Cognitive functioning (3): change scores on the Spatial pattern separation test | Baseline, post-intervention (around 6 weeks after baseline)
  The Spatial pattern separation test assesses the ability to differentiate partially overlapping patterns of activation in order to retrieve one pattern as separate from others that are similar. Specifically, it consists of 36 trials, in which the participant is required to learn the location of a grey circle on a sceen; then the participant is required to recognize the position of the previously-learned grey circle with respect to a foil located either to the left or the right of the target. Scores range from 0 to 36, where higher scores indicate better memory performance.

SECONDARY OUTCOMES:
Transfer effect on self-perceived cognitive functioning: change scores on the Subjective Memory Complaints Questionnaire | Baseline, post-intervention (around 6 weeks after baseline)
  The Subjective Memory Complaints Questionnaire assesses the subjective experience of memory decline. It consists of two sections. Part I provides a global evaluation of memory concerns responses to four general questions (4 items); Part II provides an evaluation of memory concerns in daily life (27 items). For each of the 31 items, participants are asked to respond on a 4-point Likert scale (1 = No, it does not happen to me; 2 = Sometimes, but it does not worry me; 3 = Yes and it worries me; 4 = Yes and it constitutes a problemin at least one area ofmy life, e.g., work, family, leisure, relationships). Scores range from 31 to 124. Higher scores are indicative of more serious memory complaints.
Intervention-induced changes in whole-brain functional connectivity | Baseline, post-intervention (around 6 weeks after baseline)
  Connectomics changes after intervention will be investigated between pairs of regions of the whole brain (with particular interest in areas mainly involved in training-related cognitive processes) and in the global and local topological properties of large-scale networks through graph theoretical approach.
Transfer effect on mood (1): change scores on the 30-item Geriatric Depression Scale | Baseline, post-intervention (around 6 weeks after baseline)
  It is a brief self-report questionnaire in which participants are asked to respond to the 30 questions by answering yes or no in reference to how they felt on the day of administration. Scores range from 0 to 30, where higher scores indicate higher depression.
Transfer effect on mood (2): change scores on the State-Trait Anxiety Inventory | Baseline, post-intervention (around 6 weeks after baseline)
  It is a brief self-report questionnaire to measure the presence and severity of current symptoms of anxiety and a generalized propensity to be anxious. There are two subscales within this measure: the State Anxiety Scale (S-Anxiety), which evaluates the current state of anxiety, and the Trait Anxiety Scale (T-Anxiety), which evaluates relatively stable aspects of "anxiety proneness". Range of scores for each subtest is 20-80, with higher scores indicating greater anxiety.
Transfer effect on mood (3): change scores on the 18-item Apathy Evaluation Scale (AES) | Baseline, post-intervention (around 6 weeks after baseline)
  The Apathy Evaluation Scale is a four-point Likert-Scale measure, composed of 18 items that assess and quantify emotional, behavioural and cognitive aspects of apathy. Every item is rated on a four-point response scale (0 = not at all true/characteristic to 3 = very much true/characteristic). Higher scores indicate more severe apathy.
Transfer effect on quality of life and health status: Change scores on the Short Form-36 Health Survey | Baseline, post-intervention (around 6 weeks after baseline)
  The 36-Item Health Survey taps eight health concepts, including physical functioning, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Scores range from 0 to 100, where higher scores define a more favorable health state.

CONTACTS AND LOCATIONS:
Locations (1):
- I.R.C.C.S Santa Lucia Foundation, Rome, Lazio, Italy

REFERENCES:
- [Derived] De Simone MS, Zabberoni S, Costa A, Tenaglia E, Tieri G. The effects of an immersive virtual reality and telemedicine-based multi-component intervention in individuals with subjective cognitive decline: study protocol of a randomized controlled trial. Front Psychol. 2025 Jul 11;16:1591239. doi: 10.3389/fpsyg.2025.1591239. eCollection 2025. PMID 40718565